CLINICAL TRIAL: NCT07102953
Title: The Effect of Focused Attention and Open Monitoring Meditation on Creativity in Scientific Researchers
Brief Title: Mindfulness on Creativity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Westlake University (Other); University of Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Shulin Chen, Prof., Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20250401LR001; WU2024A001 (Other Grant/Funding Number: Dingheng Shipping Technology Co. Ltd.)
Record Dates: First submitted 2025-06-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-04

CONDITIONS: Active Control; Focused-attention Meditatioin; Open-monitoring Meditation
Keywords: dismantling mindfulenss; focused-attention; open-monitoring; creativity; EEG

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focused-attention group (Experimental): Focused-attention training
  Interventions: Behavioral: Focused-attention meditation
- Open-monitoring group (Experimental): Open-monitoring training
  Interventions: Behavioral: Open-monitoring meditation
- Control group (Active Comparator): Listen to stories about creativity
  Interventions: Behavioral: Audio-listening control

INTERVENTIONS:
Behavioral: Focused-attention meditation — This is a type of mindfulenss meditation, which instructes participants to keep focusing on own breathing with a sitting and rest posture.
  Arms: Focused-attention group
Behavioral: Open-monitoring meditation — This is a type of mindfulenss meditation, which instructs participants to stay aware of their vision with a sitting and rest posture.
  Arms: Open-monitoring group
Behavioral: Audio-listening control — Participants listen to stories about creativity with a sitting and rest posture.
  Arms: Control group

SUMMARY:
Purpose of the Study

This clinical trial aims to find out whether a 5-day mindfulness training program can help improve creativity in academic researchers. The study focuses on answering these key questions:

Can focused-attention (FA) and open-monitoring (OM) meditation boost creativity in academic researchers?

Do FA and OM meditation have different effects on creativity?

How does the training affect brain activity (measured by electrical signals)?

Researchers will compare the effects of FA and OM meditation with a control group that listens to audio recordings, to see which method-if any-helps improve creativity.

What Participants Will Do

Join one of three groups: FA meditation, OM meditation, or audio listening (control), and take part in daily practice for 5 days.

Come to the research center for testing three times.

Keep a daily log of how they engage with the training.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled graduate students (Master's or PhD) or other research personnel (e.g., postdoctoral fellows, research assistants, or academic researchers).
* Aged 18 years or older and under 65 years.
* No current diagnosis of severe mental disorders (e.g., schizophrenia, schizoaffective disorder, bipolar disorder).
* Not currently taking mood-stabilizing medication (e.g., SSRIs), to avoid confounding effects on mindfulness training and EEG outcomes

Exclusion Criteria:

* Simultaneously participating in other mindfulness-based psychological intervention programs or courses that cannot be paused during the study period.
* Suicidal ideation or planning reported within the past two weeks.
* Inability to attend in-person assessments at the laboratory site.
* Refusal or inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Divergent thinking | Pre- and post- assessments after a 15-min training at Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Divergent thinking, a key component of creativity, will be assessed using the Alternative Uses Task (AUT). In this test, participants are asked to think of as many different uses as possible for a common object-like a brick, knife, or pillow-within a limited time. The scores including three factors: fluency, flexibility, and originality, which will be gained via TranDis, a semantic distance scoring system based on transformer-based language models.
Convergent thinking | Pre- and post- assessments after a 15-min training at Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Convergent thinking, a key component of creativity, will be measured by the Remote Associate Test (RAT). In this test, participants are given three words and must identify a fourth word that links all three.
EEG | During the whole tests at Day7 (after 5-day practice)
  Quantitative EEG power spectral density (PSD) across frequency bands (delta: 0.5-4 Hz, theta: 4-8 Hz, alpha: 8-13 Hz, beta: 13-30 Hz, gamma: >30 Hz) will be measured at Day 7 (post-intervention). Absolute and relative power in each band will be extracted from resting-state EEG (eyes closed), task-state EEG (15-min mindfulness or control), and task-state EEG during creativity tests, recorded at standardized scalp locations. Changes in spectral power will be used as indicators of neurophysiological responses to the mindfulness training.

SECONDARY OUTCOMES:
Mindfulness | Assessments at Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Mindfulness is assessed using the Philadelphia Mindfulness Scale (PHLMS). The PHLMS is a 20-item scale with two factors named Awareness and Acceptance. Participants will rate on a 5-point scale (1 = never, 5 = very often) according to the frequency that they experienced the described item within the past week. The score range for the PHLMS is 20 to 100.
Metacognition | At Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Cognitive Self-Consciousness (CSC), a subscale of the Metacognition Questionnaire (MCQ), will be used to assess participants' tendency to monitor and reflect upon their own thinking processes. The subscale includes 6 items. Participants rate statements such as "I am constantly aware of the way my mind works" on a 4-point scale (1 = do not agree, 5 = agree very much). The score range is 6 to 30.
Attention | Assessments at Day1 (before 5-day practice), Day7 (after 5-day practice).
  Sustained attention will be measured using the Sustained Attention to Response Task (SART). The SART is a computerized test for the measurement of sustained attention and response inhibition. Participants' performance will be evaluated by the time of response and the correct rate.
Depression | Assessments at Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 4-point scale (0 = Not at all, 3 = Nearly every day) with 9 items. The score range is 0 to 27.
Anxiety | Pre- and post- assessments after a 15-min training at Day1 (before 5-day practice), Day7 (after 5-day practice), and follow-up (1 month after 5-day practice).
  Anxiety will be measured using the Generalized Anxiety Disorder 7-item scle (GAD-7). It is a 4-point scale (0 = Not at all, 3 = Nearly every day) with 7 items. The score range is 0 to 21.

OTHER OUTCOMES:
Engagement and practice times | Day 2 to Day 5 during the intervention, and 1 month after the 5-day practice period, for participants who engaged in follow-up practice.
  Particpants will report their engagement after everyday practice by answering the question "On a scale from 0 to 10, how would you rate your level of engagement during today's practice? (0 = not engaged at all, frequent mind-wandering or drowsiness; 10 = highly engaged, focused and alert)"

CONTACTS AND LOCATIONS:
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data will be shared: demographic information, assessment scores, and time points of data collection. No personally identifiable information will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year and ending 5 years after publication
Access Criteria: Criteria for data sharing:
  Researchers must submit a scientific proposal describing the purpose and methods of the planned analyses. The analyses should be aligned with the original study objectives and must not attempt to identify individual participants. The proposal may be reviewed by the study team for scientific and ethical appropriateness.
  Mechanism for data sharing:
  Researchers need to submit a proposal and sign a data sharing agreement. Requests can be sent via email to the corresponding author. Approved researchers will receive access to the de-identified data through a secure transfer method.